CLINICAL TRIAL: NCT05634408
Title: Evaluating ACUVUE® Abiliti™ 1-Day Soft Therapeutic Lenses for Myopia Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6499
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEST Lens (Experimental): Eligible subjects will bilaterally wear the TEST Lens for the duration of the study.
  Interventions: Device: ACUVUE® Abiliti™ 1-Day Soft Therapeutic Lenses for Myopia Management (A1D)

INTERVENTIONS:
Device: ACUVUE® Abiliti™ 1-Day Soft Therapeutic Lenses for Myopia Management (A1D) — TEST Lens

SUMMARY:
This is a single-site, prospective, single-arm, open-label, real-world evidence study with a minimal study duration of 1-year, up to 2-year follow-up to evaluate overall visual acuity.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject's parents or legal guardians must read, understand, and sign the STATEMENT OF INFORMED CONSENT (Parental Permission Form and Authorization to Use and Disclose Medical Information). The subject must read (or be read to) and sign the CHILDREN'S ASSENT (Information and Assent Form) and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Between 7 and 12 (inclusive) years of age at the time of screening.
4. Be of Chinese ethnicity, which is defined as with both biological parents being of Chinese ethnicity).
5. Have normal eyes (i.e., no ocular medications or infections of any type).
6. Have non-vertex corrected subjective spherical distance refraction in the range of -0.75 D to -4.50 D (inclusive) in each eye.
7. Have refractive cylinder in the range of 0.00 D to 1.00 D (inclusive) in each eye with any degree of axis, by subjective sphero-cylindrical refraction.
8. Have sphero-cylindrical best-corrected visual acuity of 0.04 logMAR (4.95 in China standard 5-point logMAR scoring convention) or better in each eye, and the difference of sphero-cylindrical best-corrected visual acuity between the two eyes is less than 0.20 logMAR (0.2 points difference in China standard 5-point logMAR scoring convention).
9. Spherical equivalent power of cycloplegic objective spherocylindrical refraction (by auto refraction) between -0.75 D and -4.50 D (inclusive) and cylinder power of 1.00 D or less in each eye (based on the average of 5 repeated sphero-cylindrical refraction measures and rounded to the nearest 1/8 D).
10. The difference in spherical equivalent power between the two eyes be less than or equal to 1.50 D (based on the average of 5 repeated sphero-cylindrical refraction measures and rounded to the nearest 1/8 D).

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Have any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g., rheumatoid arthritis), any underlying medical condition that makes subjects at risk of severe COVID complications, or other diseases, by parent of legal guardian's self-report, which are known to interfere with contact lens wear and/or participation in the study.
2. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear and/or participation in the study. See Section 9 for additional details regarding excluded systemic medications.
3. Any current use of ocular medication (occasional use of re-wetting drops is allowed).
4. Chronic or seasonal use of ophthalmic topical medication that are specified as disallowed medications in Section 9 of the protocol.
5. Chronic use of any topical antimuscarinic agents for any reason.
6. Recent temporary use (within 21 days from enrollment) of topical agents with anti-muscarinic properties. This includes but is not limited to scopolamine, pirenzepine, tropicamide, cyclopentolate and homatropine.
7. Any known hypersensitivity or allergic reaction to cyclopentolate, topical anesthetics or Sponsor approved rewetting drop solutions available in local markets.
8. Any previous or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
9. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
10. History of myopia control treatment or participation in any prior myopia control clinical study in the test group with an optical intervention for more than 2 weeks. This includes but is not limited to orthokeratology treatment or use of other ophthalmic devices (e.g., bifocal, multifocal or other novel contact or spectacles lenses).
11. History of myopia control treatment or participation in any prior myopia control clinical study in the test group with any pharmacological intervention (e.g., atropine or pirenzepine).
12. Current or recent (within 60 days from enrollment) wear of orthokeratology lenses, bifocal, multifocal contact lenses or bifocal, multifocal spectacles.
13. Be current or recent (within 30 days from enrollment) rigid lens wearers.
14. Be immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
15. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, ocular hypertension, glaucoma, history of recurrent corneal erosions, aphakia, uveitis, severe keratoconjunctivitis sicca, keratoconus, keratoconus suspect, and pellucid marginal degeneration.
16. Grade 3 or greater palpebral conjunctival observations or any other Grade 2 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, conjunctival injection) on the ISO 11980 classification scale.
17. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear or subjects' participation in the study.
18. Any central corneal scar.
19. Any corneal distortion resulting from ocular diseases or previous hard or rigid gas permeable contact lens wear.
20. Binocular vision abnormality, intermittent strabismus or strabismus.
21. Anterior chamber angle is Grade 2 or narrower in either eye.
22. Intraocular pressure (IOP) is higher than 21 mmHg in either eye
23. Pupil diameter under bright illumination is less than 2 mm in either eye.
24. Pupil pathology.
25. Fundus pathology.
26. Any other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2022-12-24 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Change in Axial Length (AL) from baseline | Up to 24-month follow-up
  AL will be measured, in mm, every 6 months throughout the study using an ocular biometer.
Change in Spherical Equivalent of Cycloplegic Autorefraction (SECAR) from baseline | up to 24-month follow-up
  SECAR will be measured, in diopter (D), every 6 months throughout the study using an autorefractor.
Serious and significant ocular adverse events (AEs) | up to 24-month follow-up
  Number (n, %) of subjects and eyes with contact lens related (i.e., related and possibly related) serious and significant ocular adverse events (AEs) by diagnosis.

SECONDARY OUTCOMES:
Distance LogMAR Visual Acuity | up to 24-month follow-up
  Monocular and binocular distance visual acuity will be measured at distance 4 meters under high luminance (120-200 cd/m2), high contrast (>600 lux) conditions using Landolt C logMAR visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- Hainan Boao Lecheng AIER Eye Hospital Co. LTD, Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu